CLINICAL TRIAL: NCT02922439
Title: Health Literacy Assessment and Intervention to Reduce Disparities: FLIGHT/VIDAS II
Acronym: FV2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD010368
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Fatigue; Depression; Pain; Sleep Wake Disorders; Chronic Disease
Keywords: chronic disease; multimorbidity; chronic disease self-management; tailored information; mobile applications
MeSH Terms: conditions — Fatigue; Depression; Pain; Sleep Wake Disorders; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored Intervention (Experimental): Individuals will interact with a chronic disease self-management application that provides information tailored to age, race, language (English or Spanish) and level of health literacy.
  Interventions: Behavioral: Tailored Intervention
- Control (Active Comparator): Individuals will interact with a chronic disease self-management application that provides the same information as the experimental intervention but is not personally tailored to level of health literacy.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Tailored Intervention — The intervention will focus on improving the health literacy of low literacy individuals by providing chronic disease self-management information tailored to cultural and linguistic characteristics of participants.
  Arms: Tailored Intervention
Behavioral: Control Intervention — This intervention will provide information similar to that provided in the control condition, but will not utilize tailoring.
  Arms: Control

SUMMARY:
The purpose of this study will to be to evaluate the effects of a mobile intervention focused on improving the chronic disease self management skills of individuals with low health literacy. The intervention will provide information that culturally and linguistically tailored to participants' level of health literacy.

DETAILED DESCRIPTION:
Health literacy is a critically important skill that helps people to become active participants in their health care. The 2003 National Assessment of Adult Literacy showed that more than 75 million Americans had basic health literacy skills, indicating that as many as 1 in 4 Americans can have difficulty understanding information about their healthcare. Persons in racial and ethnic minorities are likely to have even lower levels of health literacy. Twenty-four percent of blacks (9.5 million persons) and 41% of Hispanics (21 million persons) have below basic levels of health literacy. These persons have lower levels of health literacy and compelling evidence, including our own findings (see below), link race and ethnicity to disparities in health via health literacy. Members of minority groups and older adults are more frequently affected by chronic diseases such as cancer, high blood pressure, heart attack, stroke, diabetes, elevated cholesterol, asthma, hepatitis C, HIV infection, mental health disorders and many others. The twin burdens of chronic disease and low levels of health literacy thus fall disproportionately on those most in need - members of minorities and older adults, all of whom likely to experience one or more chronic conditions while often not having the health literacy skills to help them cope.

Chronic disease self-management (CDSM) is a logical target for a general health literacy intervention. In an approach that cuts across specific diseases. CDSM targets problems and skills needed to cope with issues such as fatigue, pain, stress, depression, sleep disturbance and treatment adherence. Studies show that in-person CDSM classes improve patients' functioning and reduce healthcare utilization, but their availability is limited due to the lack of qualified personnel and cost. Similarly, while interventions have been developed to improve health literacy, they are difficult to scale to levels needed to meet the challenge of low health literacy (for more than 40 million persons) due to their cost. Effective interventions with the potential for wider dissemination at reasonable costs are urgently needed.

In a previous study, the investigators showed that a computer-delivered tailored information intervention targeting health literacy that can deployed either as an information kiosk in a clinical office or on the Internet could be cost-effective in improving patients' health literacy and adherence. It is not clear, however, whether the same sort of computer-delivered, multimedia and interactive approach will be effective in improving CDSM skills in persons with low baseline levels of health literacy, and if it is, whether its effects will extend beyond health literacy to general health, self-efficacy, activation, and treatment adherence. In this follow-up study the investigators will evaluate this possibility by creating a personally relevant computer-delivered intervention targeting CDSM and health literacy among African-Americans, Hispanics, and white non-Hispanics:

ELIGIBILITY:
Inclusion Criteria:

* Have at least one chronic condition (cardiovascular disease,; arthritis; cancer; lung disease, osteoporosis, depression and others treated with at least one medication
* Health literacy at or below 8th grade level as assessed by screening measure
* Able to provide informed consent

Exclusion Criteria:

* Severe cognitive disability that would preclude the ability to give informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Health Literacy | Baseline, six weeks, and three months.
  Using the FLIGHT/VIDAS health literacy scale, change in health literacy will be assessed at baseline, 6 weeks and three months.

SECONDARY OUTCOMES:
Mood | Baseline, six weeks, and three months.
  Using the Center for Epidemiological Studies Depression scale, participant mood will be assessed at baseline, six weeks and three months.
Sleep quality | Baseline, six weeks, and three months.
  Using the Insomnia Severity Index, participant sleep quality will be assessed at six weeks and three months.
Patient Activation | Baseline, six weeks, and three months.
  Using the Patient Activation Measure (scale), participant mood will be assessed at baseline, six weeks and three months.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- NSU Psychiatry Research Office -- Center for Collaborative Research, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
At study conclusion a cleaned data set will be made available to interested researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available approximately 12 months after the date of the last participant completion.
Access Criteria: Data will be made available to any interested investigator.

REFERENCES:
- [Background] Ownby RL, Acevedo A, Waldrop-Valverde D, Jacobs RJ, Caballero J, Davenport R, Homs AM, Czaja SJ, Loewenstein D. Development and initial validation of a computer-administered health literacy assessment in Spanish and English: FLIGHT/VIDAS. Patient Relat Outcome Meas. 2013 Aug 19;4:21-35. doi: 10.2147/PROM.S48384. eCollection 2013. PMID 23990736
- [Background] Ownby RL, Acevedo A, Waldrop-Valverde D, Jacobs RJ, Caballero J. Abilities, skills and knowledge in measures of health literacy. Patient Educ Couns. 2014 May;95(2):211-7. doi: 10.1016/j.pec.2014.02.002. Epub 2014 Feb 16. PMID 24637163
- [Background] Ownby RL, Acevedo A, Jacobs RJ, Caballero J, Waldrop-Valverde D. Quality of life, health status, and health service utilization related to a new measure of health literacy: FLIGHT/VIDAS. Patient Educ Couns. 2014 Sep;96(3):404-10. doi: 10.1016/j.pec.2014.05.005. Epub 2014 May 14. PMID 24856447
- [Derived] Ownby RL, Waldrop D, Davenport R, Simonson M, Caballero J, Thomas-Purcell K, Purcell D, Ayala V, Gonzalez J, Patel N, Kondwani K. A mobile app for chronic disease self-management for individuals with low health literacy: A multisite randomized controlled clinical trial. medRxiv [Preprint]. 2023 Apr 3:2023.04.01.23288020. doi: 10.1101/2023.04.01.23288020. PMID 37066256
- [Derived] Ownby RL, Acevedo A, Waldrop-Valverde D, Caballero J, Simonson M, Davenport R, Kondwani K, Jacobs RJ. A Mobile App for Chronic Disease Self-Management: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Apr 5;6(4):e53. doi: 10.2196/resprot.7272. PMID 28381395
- See also: Central study website including links to presentations and publications as well as most up-to-date information on study progress. — http://www.flightvidas.org